CLINICAL TRIAL: NCT03339063
Title: The Italian Registry of Pulmonary Non-tuberculous Mycobacteria
Acronym: IRENE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Niguarda Hospital (Other); Azienda Ospedaliera San Gerardo di Monza (Other); ASST Fatebenefratelli Sacco (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); University of Turin, Italy (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Azienda Unità Locale Socio Sanitaria n.9 Treviso (Other); Ospedale Maggiore Di Trieste (Other); Azienda Ospedaliero-Universitaria di Modena (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Università degli Studi di Ferrara (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Ospedale San Jacopo, Pistoia, Italy (Unknown); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Policlinico Umberto I (Other); Istituto Nazionale per le Malattie Infettive Spallanzani, Roma (Unknown); Policlinico Universitario, Catania (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other); Azienda Ospedaliera Cosenza (Other); Azienda Ospedaliero Universitaria di Sassari (Other)
Responsible Party: Sponsor
Other Study IDs: IRENE
Record Dates: First submitted 2017-10-22; First posted 2017-11-13 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2017-11

CONDITIONS: Nontuberculous Mycobacteria
Keywords: Nontuberculous Mycobacteria; Non-tuberculous mycobacteria; NTM-PD; NTM-LD; MAC; M. avium; M. intracellulare; M. abscessus; Atypical mycobacteria; NTM
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Sputum Bronchoalveolar lavage Full Blood Serum Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Italian registry of pulmonary non-tuberculous mycobacteria (NTM) -IRENE- is an observational, multicenter, prospective, cohort study enrolling consecutive adult patients with either a NTM respiratory infection or NTM-Pulmonary Disease. The coordinating center is located at the Pulmonary Department of the Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy. So far, more than 35 centers, including mainly pulmonary and infectious disease departments, joined the registry. The registry has been developed to accept an unlimited number of patients and no deadlines have been decided.

DETAILED DESCRIPTION:
The epidemiology of patients suffering from a pulmonary disease due to NTM (NTM-PD), which is characterized by symptomatic, progressive inflammatory lung damage and defined in 2007 in the ATS/IDSA guidelines, still remains unclear. Reporting of NTM-PD to health authorities is often not mandated in several countries and the current estimates have been obtained from sentinel surveillance or laboratory-based studies, retrospective cohort studies, or audits of administrative databases. Until now no data have been published on the epidemiology of respiratory NTM infections in Italy.

The Italian registry of pulmonary NTM (IRENE) is an observational, multicenter, prospective, cohort study enrolling consecutive adult patients with either a NTM respiratory infection or NTM-PD. The coordinating center is located at the Pulmonary Department of the Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy. So far, more than 35 centers, including mainly pulmonary and infectious disease departments, joined the registry. The study is sponsored by the Policlinico Hospital in Milan. The study website is located at www.registroirene.it.

Adult (>=18 years) patients with all of the following are included in the registry: 1) at least one positive culture for any NTM species from any respiratory sample; 2) at least one positive culture for NTM isolated in the year prior the enrolment and/or prescribed NTM treatment in the year prior the enrolment; 3) Given consent to inclusion in the study. No exclusion criteria are applied to the study. Patients included in the registry are mainly recruited among pulmonary and ID out- and in-patient services. Adult cystic fibrosis, lung transplant, and tuberculosis clinics represent other recruitment centers. The registry has been developed to accept an unlimited number of patients and no deadlines have been decided.

Patients are managed according to standard operating procedures implemented in each IRENE clinical center without any interference from the study team. A baseline case report form is collected at patient's enrolment including demographics, comorbidities, microbiological, laboratory, functional, radiological, clinical, and treatment data. Then, study investigators enter follow-up data on an annual basis.

An IRENE biobank has also been developed within the network and linked to the clinical data of the registry. IRENE sites can collect samples, including blood, serum, plasma, respiratory specimens (sputum, induced sputum, tracheal aspirate, or bronchoalveolar lavage), urine, and NTM isolates at the first visit and during follow up on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria (all of them):

* Adult (>=18 years) patients
* At least one positive culture for any NTM species from any respiratory sample
* At least one positive culture for NTM isolated in the year prior the enrolment and/or prescribed NTM treatment in the year prior the enrollment
* Given consent to inclusion in the study.

Exclusion Criteria:

No exclusion criteria are applied to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the registry are mainly recruited among pulmonary and Infectious diseases out- and in-patient services. Adult cystic fibrosis, lung transplant, and tuberculosis clinics represent other recruitment centers. A heterogeneous population of patients with NTM infection/NTM-Pulmonary Disease sharing different clinical phenotypes is expected to be enrolled in the registry. IRENE has a special focus on four patients' categories: 1) immunocompetent/bronchiectatic, 2) HIV-positive, 3) cystic fibrosis and 4) lung transplanted patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-04-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients meeting the quality standards for NTM-PD care suggested by international guidelines (including the latest ERS 2017 guidelines) | 5 years
  The number of patients with NTM-PD who have been managed or treated according to the recommendations published by international guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Aliberti, MD, Study Director — Department of Pathophysiology and Transplantation, University of Milan Internal Medicine Department, Respiratory Unit and Cystic Fibrosis Adult Center Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy; Francesco Blasi, MD, Study Chair — Department of Pathophysiology and Transplantation, University of Milan Internal Medicine Department, Respiratory Unit and Cystic Fibrosis Adult Center Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy; Luigi Ruffo Codecasa, MD, Study Chair — Regional TB Reference Centre, Istituto Villa Marelli, ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy; Andrea Gori, MD, Study Chair — Clinic of Infectious Diseases, 'San Gerardo" Hospital-ASST Monza, University Milano-Bicocca, Milano, Italy
Locations (26):
- Italy (26):
  - Clinic of Infectious Diseases, 'San Gerardo" Hospital-ASST Monza, University Milano-Bicocca, Milano, Monza, Monza Brianza
  - Malattie Infettive, Alma Mater Studiorum Università di Bologna, Bologna
  - Pneumologia, Alma Mater Studiorum Università di Bologna, Bologna
  - Clinica di Malattie Infettive e Malattie Tropicali, Spedali Civili di Brescia, Università di Brescia, Brescia
  - Malattie Infettive, Ospedale Garibaldi-NESIMA di Catania, Catania
  - U.O.C. Malattie Infettive, Azienda Ospedaliera di Cosenza, Cosenza
  - Pneumologia, Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Dipartimento Medicina Sperimentale e Clinica, SOD Malattie Infettive e Tropicali, Azienda Ospedaliero Universitaria Careggi, Florence
  - Malattie Infettive, IRCCS-AOU San Martino, Genova
  - Department of Pathophysiology and Transplantation, University of Milan Internal Medicine Department, Respiratory Unit and Cystic Fibrosis Adult Center Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Malattie Infettive, Ospedale Luigi Sacco, Milan
  - Pneumologia, Ospedale Luigi Sacco, Milan
  - Regional TB Reference Centre, Istituto Villa Marelli, ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy, Milan
  - Malattie Infettive, Ospedale di Modena, Modena
  - Pneumologia, Ospedale di Modena, Modena
  - Pneumologia, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Pneumologia, Ospedale di Pisa, Pisa
  - S.O.C. Malattie Infettive II, AUSL Toscana Centro - Pistoia, Ospedale San Jacopo, Pistoia
  - Pneumologia, Policlinico Gemelli, Roma
  - UOC di Medicina Interna e Disfunzioni Respiratorie, Azienda Universitaria Ospedaliera Policlinico Umberto I di Roma, Roma
  - UOS Day Service Malattia Tubercolare afferente all'UOC Malattie Infettive dell'Apparato Respiratorio, Istituto Nazionale per le Malattie Infettive "L. Spallanzani" - IRCCS, Roma
  - Pneumologia, Dipartimento Di Medicina Clinica e Sperimentale, Università degli studi di Sassari, Sassari
  - Divisione di Pneumologia, AOU Città della Salute e della Scienza di Torino, Molinette, Torino
  - Malattie Infettive, Università degli studi di Torino, Torino
  - UO di Pneumotisiologia, Ospedale di Vittorio Veneto, Treviso
  - Dipartimento di Pneumologia, Ospedale Universitario di Cattinara, Trieste

IPD SHARING:
Plan to Share IPD: Yes
IRENE is the official Italian network within the EMBARC European NTM registry. All Italian patients included in the European NTM registry will be enrolled through IRENE and IRENE data will be incorporated into the European NTM registry.
Supporting Information: Study Protocol
Time Frame: 2018-2023
Access Criteria: All the patients' data

REFERENCES:
- [Background] Haworth CS, Banks J, Capstick T, Fisher AJ, Gorsuch T, Laurenson IF, Leitch A, Loebinger MR, Milburn HJ, Nightingale M, Ormerod P, Shingadia D, Smith D, Whitehead N, Wilson R, Floto RA. British Thoracic Society guidelines for the management of non-tuberculous mycobacterial pulmonary disease (NTM-PD). Thorax. 2017 Nov;72(Suppl 2):ii1-ii64. doi: 10.1136/thoraxjnl-2017-210927. No abstract available. PMID 29054853
- [Background] Faverio P, Stainer A, Bonaiti G, Zucchetti SC, Simonetta E, Lapadula G, Marruchella A, Gori A, Blasi F, Codecasa L, Pesci A, Chalmers JD, Loebinger MR, Aliberti S. Characterizing Non-Tuberculous Mycobacteria Infection in Bronchiectasis. Int J Mol Sci. 2016 Nov 16;17(11):1913. doi: 10.3390/ijms17111913. PMID 27854334
- [Background] Bonaiti G, Pesci A, Marruchella A, Lapadula G, Gori A, Aliberti S. Nontuberculous Mycobacteria in Noncystic Fibrosis Bronchiectasis. Biomed Res Int. 2015;2015:197950. doi: 10.1155/2015/197950. Epub 2015 May 27. PMID 26106603
- [Background] Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. doi: 10.1164/rccm.200604-571ST. No abstract available. PMID 17277290
- [Background] Floto RA, Olivier KN, Saiman L, Daley CL, Herrmann JL, Nick JA, Noone PG, Bilton D, Corris P, Gibson RL, Hempstead SE, Koetz K, Sabadosa KA, Sermet-Gaudelus I, Smyth AR, van Ingen J, Wallace RJ, Winthrop KL, Marshall BC, Haworth CS; US Cystic Fibrosis Foundation and European Cystic Fibrosis Society. US Cystic Fibrosis Foundation and European Cystic Fibrosis Society consensus recommendations for the management of non-tuberculous mycobacteria in individuals with cystic fibrosis. Thorax. 2016 Jan;71 Suppl 1(Suppl 1):i1-22. doi: 10.1136/thoraxjnl-2015-207360. PMID 26666259
- [Derived] Aliberti S, Codecasa LR, Gori A, Sotgiu G, Spotti M, Di Biagio A, Calcagno A, Nardini S, Assael BM, Tortoli E, Besozzi G, Ferrarese M, Matteelli A, Girardi E, De Lorenzo S, Seia M, Gramegna A, Del Prato B, Terranova L, Oriano M, Sverzellati N, Mirsaeidi M, Chalmers JD, Haworth CS, Loebinger MR, Aksamit T, Winthrop K, Ringshausen FC, Previdi G, Blasi F; IRENE Network. The Italian registry of pulmonary non-tuberculous mycobacteria - IRENE: the study protocol. Multidiscip Respir Med. 2018 Aug 9;13(Suppl 1):33. doi: 10.1186/s40248-018-0141-8. eCollection 2018. PMID 30151192

DOCUMENTS (2):
  • Study Protocol (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT03339063/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT03339063/SAP_001.pdf